CLINICAL TRIAL: NCT00435006
Title: Hypopituitarism Following Traumatic Brain Injury or Spontaneous Subarachnoidal Haemorrhages
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Novo Nordisk A/S (Industry); AP Moeller Foundation (Other)
Other Study IDs: KF-01-107/03
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2007-02-14 (Estimated); Status verified 2007-02

CONDITIONS: Brain Injuries; Intracranial Aneurysm
MeSH Terms: conditions — Brain Injuries; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to assess the prevalence and predictors of pituitary dysfunction, as well as secondary out-come in patients with traumatic brain injury or spontaneous subarachnoidal haemorrhages.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of traumatic brain injury (TBI) or subarachnoidal haemorrhages (SAH)

Exclusion Criteria:

* Alcohol or drug abuse
* Prior TBI or SAH
* Chronic use of glucocorticoids
* Pregnancy or breast feeding
* Diagnosis of psychiatric diseases or malignant neoplasms

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Marianne C Klose, MD, Principal Investigator — Dept. of Endocrinology PE2131, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Dept. of Endocrinology PE2131, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark